CLINICAL TRIAL: NCT02464813
Title: Effect of Pregabalin on Immediate Post-operative and Longterm Pain and Spinal Cord Monitoring in Children Undergoing Instrumented Spinal Surgery.
Brief Title: Effect of Pregabalin on Immediate Post-operative and Longterm Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Ilkka Helenius, Division Head, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: T93/2015; 2015-000072-99 (EudraCT Number)
Record Dates: First submitted 2015-05-15; First posted 2015-06-08 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Scoliosis; Spondylolisthesis
Keywords: pregabalin; idiopathic scoliosis
MeSH Terms: conditions — Scoliosis; Spondylolisthesis | interventions — Pregabalin; Sugars; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregabalin (Active Comparator): Pregabalin in hard capsule 2mg/kg rounded up to next 25mg twice daily, max 150mg x 2, for 5 days.
  Interventions: Drug: Pregabalin; Drug: Oxycodone
- Sugar pill (Placebo Comparator): Same hard capsule and same amount of tablets twice daily for 5 days.
  Interventions: Drug: Sugar pill; Drug: Oxycodone

INTERVENTIONS:
Drug: Pregabalin — Patients will receive pregabalin twice preoperatively and twice daily for 5 days after surgery.
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Sugar pill — Patients will receive placebo twice preoperatively and twice daily for 5 days after surgery.
  Other Names: placebo
  Arms: Sugar pill
Drug: Oxycodone — All patients will receive oxycodone as analgetic treatment administered by PCA. Oxycodone consumption will be measured.

SUMMARY:
This study aims to evaluate the incidence of longterm pain after spinal fusion surgery in children and adolescents. In the second part of the study a randomized double-blind clinical trial will be conducted. We compare the effect of pregabalin versus placebo on postoperative pain and oxycodone consumption. We will also be able to evaluate the effect of pregabalin on neurophysiological monitoring during surgery.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis is the most common indication for major surgery during adolescence. Postoperative pain is a major concern in these adolescents with major surgical trauma. Spinal cord monitoring is an essential part of spinal deformity correction, but the effects of pregabalin on these measurements are not known.

In order to evaluate the incidence of longterm postoperative pain in children after spinal surgery the first part of our study will be retrospective. We will send a symptom and pain questionnaire to all children, who have been in spinal fusion surgery at our university hospital between the years 2009-2015. The questionnaire will include Oswestry Low Back Pain Questionnaire, pain drawing and SRS-24. The Oswestry Disability Index is currently considered by many as the gold standard for measuring degree of disability and estimating quality of life in a person with low back pain.

In the second part of our study a randomized double-blind clinical trial will be conducted comparing the effect of pregabalin and placebo on postoperative pain and oxycodone consumption. In addition the effect of pregabalin on neurophysiological monitoring in adolescents undergoing surgery for spinal deformities will be assessed. Finally, the prevalence of persistent postsurgical pain will be evaluated at 6, 12 and 24 months after surgery.

To obtain statistical power of 80% and a type I-error level of 0.05, 60 adolescents (30 in control and 30 in active treatment group) will be recruited according to CONSORT guidelines.

The aim of the study is to evaluate the effect of pregabalin given twice preoperatively and for five days postoperatively on postoperative pain. Pain will be measured using visual analogue scale (VAS). Oxycodone administered using patient controlled anesthesia (PCA) will be used for analgesia. Persistent pain at 6, 12 and 24 months will also be evaluated. In addition, the effect of preoperative pregabalin on motor evoked potentials (latency, amplitude, currency needed to evoke potentials) during spinal cord monitoring as well as perioperative EEG findings and on the consumption of anesthetics.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent (10-21 years) undergoing spinal fusion for idiopathic scoliosis, spondylolisthesis or Scheuermann kyphosis.
2. Posterior spinal fusion
3. No contraindication for Pregabalin use
4. ASA I-III
5. Written informed consent

Exclusion Criteria:

1. Other spinal pathology or other associated medical condition
2. Major neurologic developmental delay
3. Need for anterior surgery or for vertebral column resection.
4. Preoperative opioid use
5. Inability to use PCA

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain measured in oxycodone consumption | 0-48h postoperatively
  All patients will receive oxycodone as analgesia administered using PCA. The oxycodone consumption will be recorded every 8 h. All adverse effects will be recorded. The oxycodone consumption will be measured in mg/kg/d.

SECONDARY OUTCOMES:
Effect on neurophysiological measurements during spinal surgery | First 24 h.
  As a golden standard motor evoked potentials will be recorded and measured during surgery. The latency, amplitude and currency needed to evoke the potentials will be recorded.
Effect on incidence of longterm pain | 2 years after surgery
  At the 2 year follow-up the patients will answer a pain questionnaire, Oswestry Low Back Pain Questionnaire and a pain drawing. The incidence of longterm pain after surgery will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland